CLINICAL TRIAL: NCT01893502
Title: Smoke Free Randomized Controlled Trial
Brief Title: Duration of Follow-Up Counselling on Smoking Cessation Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Dr. See Kay Choong, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/00057
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Participants will receive weekly proactive and live telephone counselling from Quitline (run by the Health Promotion Board) for one month
  Interventions: Behavioral: Telephone counselling from Quitline
- Group 2 (Active Comparator): Participants will receive weekly proactive and live telephone counselling from Quitline (run by the Health Promotion Board) for six months
  Interventions: Behavioral: Telephone counselling from Quitline

INTERVENTIONS:
Behavioral: Telephone counselling from Quitline

SUMMARY:
Smoking cessation improves mortality, even in patients with existing smoking-related morbidity. Telephone follow-up after smoking cessation counselling as been shown to be an important method to provide support to smokers and to improve quit rates, especially if three or more calls were used in addition to face-to-face counselling. While it is reasonable to assume that more counselling leads to better smoking cessation outcomes, little evidence exists over the amount of telephone follow-up counselling that is required for optimal and sustained abstinence. We aim to investigate if six-months of weekly telephone follow-up is superior to one-month of weekly telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers among outpatients, including hospital employees, who provide informed consent for enrollment in the smoking cessation program

Exclusion Criteria:

* Subjects who decline smoking cessation or who do not provide informed consent
* Subjects who are participating or will be participating in other smoking cessation programs within the next six months
* Subjects who are currently using smoking cessation medications
* Subjects who cannot be followed up for at least six months, for instance, subjects who would be resigning and going overseas within the next six months
* Subjects with language limitations that would impede completion of self-administered questionnaires
* Subjects who are difficult to communicate with over the telephone (e.g. having speech or hearing problems)
* Subjects with cognitive impairments that would impede counselling and follow-up
* Subjects with no telephone number
* Subjects who are too sick to receive smoking cessation counselling
* Subjects with limited life expectancy (e.g. metastatic cancer)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

PRIMARY OUTCOMES:
Seven-day point prevalence abstinence | Six months

SECONDARY OUTCOMES:
Average number of cigarettes smoked per day over the past seven days | 3, 6, 12 months

OTHER OUTCOMES:
Exhaled carbon monoxide levels | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kay C See, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore